CLINICAL TRIAL: NCT06085898
Title: Assessment of Dermal Acceptance, Gynecological and pH Maintenance With Microbiological Analysis of Vaginal Secretion for Cosmetic Product
Brief Title: Stryphnodendron Adstringens Intimate Soap
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Biolab Sanus Farmaceutica (Industry)
Collaborators: Medcin Instituto da Pele (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EN22-0629-01
Record Dates: First submitted 2023-07-06; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Vaginal Flora Imbalance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stryphnodendron Adstringens (Barbatimão) (Experimental): Intimate Soap
  Interventions: Drug: Stryphnodendron Adstringens 3% - once daily post bath

INTERVENTIONS:
Drug: Stryphnodendron Adstringens 3% - once daily post bath — Intimate Soap
  Other Names: Barbatimão

SUMMARY:
This is a single-centre, single-blind, non-comparative clinical trial to assess the safety of the investigational product through clinical probability assessment.

Thirty-three female participants, aged between 18-45, will be required. Assessment of dermal (dermatological) and gynecological acceptance, in addition to pH measurements and vaginal force collection for microbiological analysis at the beginning and end of the study.

DETAILED DESCRIPTION:
This is a single-centre, single-blind, non-comparative clinical trial to assess the safety of the investigational product through clinical probability assessment.

Thirty-three female participants, aged between 18-45, will be required. Assessment of dermal (dermatological) and gynecological acceptance, in addition to pH measurements and vaginal force collection for microbiological analysis at the beginning and end of the study.

Participants will remain in the study for a minimum period of 30 days, using the product for the same period according to the flow below:

Flow of Visits:

Visit 01 (D0)

* Participants' consent process after understanding the study;
* Initial assessments: safety clinics (dermatologist/gynecologist);
* Vaginal pH measurement;
* Collection of vaginal secretion;
* Dispensing of the usage diary;
* Investigational product dispensing.

Visit 02 (D30 ±2 days)

* Final assessments: clinical safety assessments (dermatologist/gynecologist);
* Vaginal pH measurement;
* Collection of vaginal secretion;
* Collection of the usage diary;
* Return of the product;
* Subjective questionnaire (self-assessment) to capture possible feelings of discomfort;
* Completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Active and regular menstrual flow;
* Vaginal pH value between 3.8 and 4.5;
* Intact skin in the product analysis region (vaginal mucosa);
* Being a user of cosmetic products of the same category (intimate soap);
* Agreement to follow the trial procedures and attendance at the Clinical Research Center on the days and times determined for applications and/or estimates;
* Understanding, consent and signature of the Free and Informed Consent Term (TCLE).

Exclusion Criteria:

* Participants who have been diagnosed with COVID-19 in the last 4 weeks or who have symptoms such as fever, dry cough, tiredness, body aches or other discomforts;
* Pregnancy or risk of pregnancy and/or lactation;
* Being in the menstrual period;
* Use of anti-inflammatory/immunosuppressive/antihistamine drugs up to 3 weeks before selection;
* Skin marks in the experimental area that interfere with the evaluation of possible skin reactions (vascular malformations, scars, increased hairiness, large amounts of nevus, sunburn);
* Atopic or allergic history to cosmetic products;
* Pathologies and/or active skin lesions (local and/or disseminated) in the evaluation area;
* Immunosuppression by drugs or active diseases;
* Decompensated endocrinopathies;
* Relevant medical history or current evidence of alcohol or other drug abuse;
* Known history or suspected intolerance to products of the same category;
* Aesthetic or dermatological treatment in the evaluation area up to 04 weeks before selection;
* Employees of Medcin or the sponsoring company involved in the study, or a close family member of an employee involved in the study;
* Other conditions considered by the researcher as reasonable for disqualification from participation in the study. If yes, it should be described in observation in the clinical record.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-11-05 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Dermatological and gynecological evaluation criteria | Immediately after the intervention
  Assess the presence of any clinical signs/symptoms in the vulva, anal and vaginal region by visually observing the mons pubis, labia majora, labia minora, clitoris, vaginal vestibule, urethral orifice, perineum and anal region, with application of a 2-point categorical scale (0=no, 1=yes)

SECONDARY OUTCOMES:
Assessment | Assessment of the occurrence and intensity of erythema, edema, scaling and vesiculation, using a 4-point scale (0=absent, 1=mild, 2=moderate, 3=severe)
  Clinical signs and/or symptoms of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Medcin Instituto da Pele, Osasco, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No